CLINICAL TRIAL: NCT00325559
Title: The Effect of Hyperglycaemia on Local Energy Stores in the Working Muscle in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1122
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 1; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

INTERVENTIONS:
Procedure: Normoinsulinemic eu- or hyperglycemic clamp

SUMMARY:
This study aims at investigating the effect of hyperglycaemia on physical performance and local energy stores in the muscle in patients with type 1 diabetes mellitus under exercise conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged from 20 to 40 years
* Patients with type 1 diabetes mellitus lasting for at least 5 years (C-Peptide ≤ 0.3 nmol/l in the presence of a plasma glucose level ≥ 7 mmol/L, indicating insulin dependence)
* Insulin delivery by CSII (continuous subcutaneous insulin infusion) for at least 6 months
* Acceptable to good metabolic control, reflected by an HbA1c 5-8%
* Normal insulin sensitivity, reflected by a daily insulin requirement of 0.3-1.0 U/kg body weight
* minimum 30' of moderate exercise 3 times per week
* BMI in the range of 18-25 kg/m2

Exclusion Criteria:

* Chronic complications of diabetes:

  * Microalbuminuria (Mogensen nephropathy stadium ≥ III)
  * Sensory neuropathy (vibration better than 5/8 at the metatarsophalangeal articulation of digitus I)
  * Proliferating retinopathy
  * No history of macro-vascular complications
  * Clinically relevant autonomous neuropathy
* Smoking
* Abnormal thyroid function
* Major depression, psychosis and other severe personality disorders, claustrophobia
* Active neoplasia
* Contraindications to exposure to a 1.5 T magnetic field (pace-makers, osteosynthetic material, etc.)
* Abnormal liver or renal function (creatinine > 130 µmol/L; ASAT and ALAT > 3 times the upper reference limit)
* Excessive alcohol consumption (>60g/d) or drug-abuse
* Refusal to give written informed consent
* Participation in another study
* Patients, who are not suitable for the study according to the study physician

Ages: 20 Years to 40 Years | Sex: Male
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Paired difference in the time to complete a time trial corresponding to 5 km cycling between euglycaemia and hyperglycaemia

SECONDARY OUTCOMES:
Muscle glycogen content during exercise in the working muscle (pre test vs. post test), in euglycaemia and hyperglycaemia respectively (All following endpoints are paired differences (euglycaemia vs. hyperglycaemia) of paired differences (pre
IMCL content during exercise in the working muscle
Rate of appearance of glucose
Rate of disappearance of glucose
Rate of glucose infusion
Total glucose oxidation
Oxidation of endogenous glucose
Oxidation of exogenous glucose
Fat oxidation (calculated via tracer and via RER)
Rate of perceived exertion
Serum lactate levels during the exercise test
Amino acid oxidation
Serum free fatty acid concentration
Serum insulin levels
Serum glucose levels
Time to achieve hyperglycemia during clamp
Pretest diary data

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, MD, Principal Investigator — University hospital of Bern
Locations (1):
- Department of Endocrinology, Diabetes and Clinical Nutrition, University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Jenni S, Oetliker C, Allemann S, Ith M, Tappy L, Wuerth S, Egger A, Boesch C, Schneiter P, Diem P, Christ E, Stettler C. Fuel metabolism during exercise in euglycaemia and hyperglycaemia in patients with type 1 diabetes mellitus--a prospective single-blinded randomised crossover trial. Diabetologia. 2008 Aug;51(8):1457-65. doi: 10.1007/s00125-008-1045-5. Epub 2008 May 30. PMID 18512043